CLINICAL TRIAL: NCT00430235
Title: A Phase II Study of BAY 43-9006 in Combination With Bicalutamide in Patients With Chemo-Naïve Hormone Refractory Prostate Cancer
Brief Title: A Study of BAY 43-9006 in Combination With Bicalutamide in Patients With Chemo-Naïve Hormone Refractory Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Dr Kim Chi, BC Cancer Agency
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OZM-001
Record Dates: First submitted 2007-01-30; First posted 2007-02-01 (Estimated); Last update posted 2010-08-05 (Estimated); Status verified 2010-08

CONDITIONS: Adenocarcinoma of the Prostate
Keywords: prostate; cancer; BAY 43-9006
MeSH Terms: conditions — Neoplasms | interventions — Sorafenib

INTERVENTIONS:
Drug: BAY 43-9006 — BAY 43-9006, 400 mg, PO, BID in a 28-day cycle(morning and evening) Bicalutamide 50 mg po Once daily in a 28-day cycle (morning)

SUMMARY:
Purpose:

To determine the efficacy of BAY 43-9006 in combination with bicalutamide in patients with chemo-naïve hormone-refractory prostate cancer.

Hypothesis:

That there will be PSA response when BAY 43-9006 in combination with bicalutamide is given to patients with chemo-naïve hormone-refractory prostate cancer.

DETAILED DESCRIPTION:
Justification:

The biologic and clinical activity and tolerability of BAY 43-9006, the therapeutic needs of the proposed patient population, and the experimental evidence in support of targeting the VEGF/VEGFR and MAPK pathways in combination with androgen receptor blockade in prostate cancer, provides a strong rationale for the proposed phase II trial to evaluate the tolerability and anti-cancer activity of combined treatment with the non-steroidal anti-androgen bicalutamide with the multi-targeted kinase inhibitor BAY 43-9006 in patients with prostate cancer that is progressing after castration therapy.

Objectives:

The primary study objective is to define the efficacy (i.e. post treatment decrement in PSA (PSA response)) of BAY 43-9006 in combination with bicalutamide in patients with chemo-naïve hormone-refractory prostate cancer.

Secondary Objectives:

* To determine the safety and tolerability of BAY 43-9006 given in combination with bicalutamide in patients with HRPC.
* To determine the time to treatment failure, PSA progression and disease progression in HRPC patients treated with BAY 43-9006 in combination with bicalutamide.
* To determine objective response rates in HRPC patients with measurable disease treated with BAY 43-9006 in combination with bicalutamide.

Research Method:

This is a phase II clinical trial in patients with androgen independent prostate cancer which will evaluate the therapeutic activity and safety profile of BAY 43-9006 given orally at the recommended phase II dose of 400 mg PO BID continuously in combination with bicalutamide 50 mg PO daily continuously. Each 4 week period will be considered 1 cycle. Doses will be adjusted for toxicity.

Statistical Analysis:

Primary Endpoint The primary endpoint for this study will be the rate of PSA-response of the combination for patients with rising PSA post castration therapy.

Secondary Endpoints:

Secondary endpoints will include time to treatment failure, time to PSA progression, duration of PSA response, median survival time, 1 year survival rate, objective tumor response rate and stable disease rate as defined by the RECIST criteria, response duration, and incidence of toxicities by NCI CTCAE.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a histologic or cytologic diagnosis of adenocarcinoma of the prostate.
2. Patients must have low-bulk asymptomatic metastatic or biochemical recurrent disease for which no curative therapy exists.
3. Patients must have documented evidence of PSA progression while receiving androgen ablative therapy, i.e. must be hormone refractory.
4. The PSA must be > 5 μg/L at the time of study entry.
5. ECOG performance status of 0 or 1.
6. Age 18 years of age or older
7. Patients must have a life expectancy of at least 12 weeks.
8. Chemotherapy: No prior cytotoxic chemotherapy is permissible. Neoadjuvant or adjuvant chemotherapy is permissible provided it was > 12 months prior to registration.
9. Hormonal Therapy:

   * Prior hormone therapy in the form of medical or surgical castration is required. Patients must be hormone refractory and have been previously and currently treated with androgen ablative therapy.
   * Patients may have received up to one line of non-steroidal anti- androgens in combination with chemical or surgical castration. Use of prior Bicalutamide is restricted to less than 3 months of continuous usage. Patients must be off anti-androgens for at least 6 weeks prior to study entry.
10. Radiation: Prior external beam radiation is permitted provided a minimum of 4 weeks has elapsed between the last dose and enrollment to the trial.
11. Steroids. Current treatment with steroids ≤ an equivalent of prednisone 20 mg day is permitted.
12. Men of childbearing potential must use an effective form of contraception i.e. double barrier method.
13. Laboratory Requirements - within 7 days prior to enrollment Hematology: Hemoglobin ≥ 100g/L Neutrophils > 1.5 x 109/L Platelets > 100 x 109/L INR ≤ 1.5 x upper limit of normal Biochemistry: AST, ALT within normal limits Bilirubin within normal limits Serum creatinine ≤1.5 x upper limit of normal

15. Patient consent must be obtained 16. Patients must be accessible for treatment and follow-up. 17. Protocol treatment is to begin within 5 working days of patient registration.

Exclusion Criteria:

1. Prior use of BAY 43-9006 or other VEGF/VEGFR or EGFR targeting agents.
2. Patients with a history of other malignancies, except: adequately treated non-melanoma skin cancer or other solid tumours curatively treated with no evidence of disease for > 5 years.
3. Patients with known brain metastases or leptomeningeal disease
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to BAY 43-9006 or other agents used in the study.
5. Other serious intercurrent illness or medical condition that might be aggravated by protocol treatment including:myocardial infarction within 6 months prior to study entry:

   * myocardial infarction within 6 months prior to study entry
   * congestive heart failure
   * unstable angina
   * cardiomyopathy
   * unstable ventricular arrhythmia
   * uncontrolled hypertension (systolic blood pressure ≥ 160, diastolic blood pressure ≥100)
   * controlled psychotic disorders
   * serious infections
   * peptic ulcer disease
   * history of bleeding diathesis
6. Upper gastrointestinal or other conditions that would preclude compliance with oral medication.
7. Patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy. Therefore, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with BAY 43-9006. Appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated.
8. Patients who require large amounts of narcotic therapy to control pain (e.g. morphine equivalent dose > 30 mg/day) since these patients would more appropriately be offered systemic chemotherapy.
9. Patients who require therapeutic anticoagulation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2007-03; Primary Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
rate of PSA-response

SECONDARY OUTCOMES:
time to treatment failure
time to PSA progression
duration of PSA response
median survival time
1 year survival rate
objective tumor response rate
stable disease rate as defined by the RECIST criteria,
response duration
incidence of toxicities by NCI CTCAE.

CONTACTS AND LOCATIONS:
Overall Officials: Kim N Chi, MD, Study Chair — British Columbia Cancer Agency
Locations (1):
- BC Cancer Agency - Vancouver Centre, Vancouver, British Columbia, Canada